CLINICAL TRIAL: NCT04473027
Title: BLood Groups as Biomarker to Optimize Odds of Response to Anti-PD-1 Drugs (BLOOD Trial)
Brief Title: BLood Groups as Biomarker to Optimize Odds of Response to Anti-PD-1 Drugs
Acronym: BLOOD
Status: Terminated | Type: Observational
Why Stopped: Low patient inclusion
Sponsor: University Hospital, Ghent (Other)
Collaborators: Jessa Hospital (Other); University Hospital, Antwerp (Other); Algemeen Ziekenhuis Maria Middelares (Other); GZA Ziekenhuizen Campus Sint-Augustinus (Other); AZ Sint-Jan AV (Other); AZ Nikolaas (Other); AZ Sint-Lucas Gent (Other); AZ Sint-Lucas Brugge (Other); General Hospital Groeninge (Other); OLV van Lourdes Hospital Waregem (Unknown); AZ Damiaan (Unknown); AZ Delta (Other); ASZ Aalst (Other); Belgian Red Cross (Other)
Responsible Party: Sponsor
Other Study IDs: BC-5765
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2020-07

CONDITIONS: Melanoma; Cancer
Keywords: Immunotherapy; Anti-PD-1; Nivolumab; Pembrolizumab; Biomarker
MeSH Terms: conditions — Melanoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — EDTA blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with advanced melanoma: Patients receiving anti-PD-1 monotherapy (Nivolumab or Pembrolizumab) in the first-line setting
  Interventions: Diagnostic Test: Blood sample collection

INTERVENTIONS:
Diagnostic Test: Blood sample collection — Whole venous blood of participants will be collected in EDTA tubes (max. 10 mL) at baseline, before start of first immunotherapy round. The Belgian Red Cross will perform serological blood group diagnostics, and molecular RBC typing.

SUMMARY:
BLOOD is an investigator-initiated, multicenter, prospective biomarker study in patients with advanced melanoma treated with anti-PD-1 monotherapy in the first-line setting. The "studied products" will be administered and managed within routine medical care in Belgium. The overall goal is (i) to investigate biomarkers for anti-PD-1 monotherapy and (ii) to gather evidence on real-life use of anti-PD-1 monotherapy in melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven advanced melanoma.
* Anti-PD-1 monotherapy of advanced (unresectable or metastatic) melanoma (prescribed within its approved indication as per usual practice according to RIZIV/INAMI regulations) in the first-line setting.
* No prior systemic therapy for advanced melanoma.
* Have measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
* At least 18 years of age.

Exclusion Criteria:

* Prior treatment with any drug specifically targeting T-cell co-stimulation or immune checkpoints (e.g., antibodies targeting PD-(L)1 or CTLA-4, chimeric antigen receptor T (CAR-T) cell therapy).
* Metastasis-directed therapy (surgery or radiotherapy) with definitive intent (local therapy to address symptomatic sites of disease is permitted).
* Previous systemic treatment for advanced melanoma.
* Active central nervous system (CNS) metastases (previously treated brain metastases are permitted if stable) or carcinomatous meningitis.
* Diagnosis of any other malignancy within 5 years prior to study inclusion, except for adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the breast or of the cervix, low-risk prostate cancer on surveillance without any plans for treatment intervention, or prostate cancer that has been adequately treated with prostatectomy or radiotherapy and currently with no evidence of disease and symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced melanoma
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
The association between ABO blood groups (specifically O vs A/B/AB) and anti-PD-1 monotherapy efficacy. | 25 weeks
  In terms of objective response rate (ORR) according to RECIST v1.1
Descriptive data on real-life use of anti-PD-1 therapy. | 3, 6, 12 months
  Based on demographics (age, ethnicity, sex, height, weight (and Body Mass Index), smoking status, and gravida/para/abortus (if female)), melanoma history, clinical profile of participant at time of anti-PD-1 initiation, prior and/or concomitant intervention(s), duration of treatment exposure during the study, and effectiveness and safety of anti-PD-1 therapy.

SECONDARY OUTCOMES:
The association between ABO blood groups and anti-PD-1 monotherapy efficacy. | 12, 25 weeks
  In terms of Overall Response Rate (ORR) / Disease Control Rate (DCR) / Best Overall Response (BOR) (RECIST v1.1)
The association between ABO blood groups and anti-PD-1 monotherapy efficacy. | 3, 6, 12 months
  in terms of Progression-Free Survival (PFS) / Overall Survival (OS) (RECIST v1.1)
The association between Kell, Kidd, Duffy, MNS, Rhesus, and Dombrock blood group antigens and anti-PD-1 monotherapy efficacy. | 12, 25 weeks
  In terms of ORR/DCR/BOR (RECIST v1.1)
The association between Kell, Kidd, Duffy, MNS, Rhesus, and Dombrock blood group antigens and anti-PD-1 monotherapy efficacy. | 3, 6, 12 months
  In terms of PFS/OS (RECIST v1.1)
The association between irregular antibodies and anti-PD-1 monotherapy efficacy. | 12, 25 weeks
  In terms of ORR/DCR/BOR (RECIST v1.1)
The association between irregular antibodies and anti-PD-1 monotherapy efficacy. | 3, 6, 12 months
  In terms of PFS/OS (RECIST v1.1)
To evaluate the association between overall survival and other endpoints as defined in the primary endpoints. | 12 months
  (i.e., ORR, DCR, BOR, and PFS)
The association between steroid administration and anti-PD-1 monotherapy efficacy. | 12, 25 weeks
  In terms of ORR/DCR/BOR (RECIST v1.1)
The association between steroid administration and anti-PD-1 monotherapy efficacy. | 3, 6, 12 months
  In terms of PFS/OS (RECIST v1.1)
The association between immunosuppressant administration and anti-PD-1 monotherapy efficacy. | 12, 25 weeks
  In terms of ORR/DCR/BOR (RECIST v1.1)
The association between immunosuppressant administration and anti-PD-1 monotherapy efficacy. | 3, 6, 12 months
  In terms of PFS/OS (RECIST v1.1)
The association between antibiotics administration and anti-PD-1 monotherapy efficacy. | 12, 25 weeks
  In terms of ORR/DCR/BOR (RECIST v1.1)
The association between antibiotics administration and anti-PD-1 monotherapy efficacy. | 3, 6, 12 months
  In terms of PFS/OS (RECIST v1.1)
The association between selected baseline and intermediate data (as listed in Outcome 2) and anti-PD-1 monotherapy efficacy. | 12, 25 weeks
  In terms of ORR/DCR/BOR (RECIST v1.1)
The association between selected baseline and intermediate data (as listed in Outcome 2) and anti-PD-1 monotherapy efficacy. | 3, 6, 12 months
  In terms of PFS/OS (RECIST v1.1)

OTHER OUTCOMES:
The relationship between anti-PD-1 monotherapy efficacy and red blood cell transfusions. | 12, 25 weeks and 3, 6, 12 months
  In terms of ORR/DCR/BOR/PFS/OS (RECIST v1.1)
The relationship between anti-PD-1 monotherapy efficacy and vaccinations. | 12, 25 weeks and 3, 6, 12 months
  In terms of ORR/DCR/BOR/PFS/OS (RECIST v1.1)
The relationship between anti-PD-1 monotherapy efficacy and previous pregnancies. | 12, 25 weeks and 3, 6, 12 months
  In terms of ORR/DCR/BOR/PFS/OS (RECIST v1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Hannelore Denys, MD, PhD, Principal Investigator — Medical Oncologist; Emiel De Jaeghere, MD, Study Chair — PhD Fellow
Locations (1):
- University Hospital Gent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No